CLINICAL TRIAL: NCT00159770
Title: Tolerability, Safety, And Efficacy Of Ziprasidone (80 - 160 Mg/D) Versus Olanzapine (10 - 20 Mg/D), Risperidone (4 - 8 Mg/D) Or Quetiapine (300 - 750 Mg/D) In Pretreated Patients With Schizophrenia, Schizoaffective Disorder Or Schizophreniform Disorders - A 12-Week Open-Label, Multicenter Clinical Trial.
Brief Title: Effect And Safety Of Ziprasidone Compared To Other Atypical Antipsychotic Drug In Schizophrenic Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A1281079
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Psychotic Disorders
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Risperidone; Quetiapine Fumarate; Hematologic Tests

INTERVENTIONS:
Drug: ziprasidone versus olanzapine , risperidone or quetiapine
Behavioral: Panss , CGI-C, UKU-SERS-Pa
Procedure: Blood tests

SUMMARY:
Evaluation of the antipsychotic efficacy and safety of ziprasidone versus olanzapine, risperidone or quetiapine in patients with schizophrenia, schizoaffective and schizophreniform disorders under naturalistic conditions of clinical practice

ELIGIBILITY:
Inclusion Criteria:

* Inpatients or outpatients with schizophrenia, schizoaffective and schizophreniform disorders (DSM-IV).
* Patients without adequate current treatment (i.e. intolerance to their current treatment or lack of efficacy of current treatment) based on clinical judgement of the investigator

Exclusion Criteria:

* A history of intolerance to ziprasidone, olanzapine, risperidone or quetiapine or any of its ingredients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290
Dates: Start 2001-11; Study Completion 2004-09

PRIMARY OUTCOMES:
PANSS (The Positive And Negative Syndrome Scale) in a 12 week period

SECONDARY OUTCOMES:
CGI-C score (Clinical Global Impression of Change), UKU-SERS-Pa (Patient self rating version). Safety and tolerability: ECG, serum cholesterol, triglycerides, prolactin, glucose and body weight

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (43):
- Denmark (22):
  - Pfizer Investigational Site, Aalborg
  - Pfizer Investigational Site, Arhus C
  - Pfizer Investigational Site, Augustenborg
  - Pfizer Investigational Site, Ballerup Municipality
  - Pfizer Investigational Site, Brovst
  - Pfizer Investigational Site, Copenhagen
  - Pfizer Investigational Site, Dianalund
  - Pfizer Investigational Site, Esbjerg
  - Pfizer Investigational Site, Esbjerg N
  - Pfizer Investigational Site, Glostrup Municipality
  - Pfizer Investigational Site, Haderslev
  - Pfizer Investigational Site, Holbæk
  - Pfizer Investigational Site, Kjellerup
  - Pfizer Investigational Site, Kolding
  - Pfizer Investigational Site, København S
  - Pfizer Investigational Site, Lemvig
  - Pfizer Investigational Site, Odense C
  - Pfizer Investigational Site, Ringkøbing
  - Pfizer Investigational Site, Risskov
  - Pfizer Investigational Site, Vejle
  - Pfizer Investigational Site, Viborg
  - Pfizer Investigational Site, Vordingborg
- Finland (7):
  - Pfizer Investigational Site, Forssa
  - Pfizer Investigational Site, Helsinki
  - Pfizer Investigational Site, Jarvenpaa
  - Pfizer Investigational Site, Kiviranta
  - Pfizer Investigational Site, Mikkeli
  - Pfizer Investigational Site, Turku
  - Pfizer Investigational Site, Tuusula
- Pfizer Investigational Site, Reykjavik, Iceland
- Switzerland (13):
  - Pfizer Investigational Site, Basel, Canton of Basel-City
  - Pfizer Investigational Site, Bern, Canton of Bern
  - Pfizer Investigational Site, Sankt Gallen, Canton of St. Gallen
  - Pfizer Investigational Site, Lausanne, Canton of Vaud
  - Pfizer Investigational Site, Prangins, Canton of Vaud
  - Pfizer Investigational Site, Zurich, Canton of Zurich
  - Pfizer Investigational Site, Bulle
  - Pfizer Investigational Site, Chêne-Bourg
  - Pfizer Investigational Site, Delémont
  - Pfizer Investigational Site, Oetwil
  - Pfizer Investigational Site, Riehen
  - Pfizer Investigational Site, Saint Urban
  - Pfizer Investigational Site, Solothurn